CLINICAL TRIAL: NCT05634304
Title: MyOsteoarthritisMyWay: Needs Exploring, Program Developing, and Implementing of a Patient-Centered Mobile App Self-Management Program for Osteoarthritis
Brief Title: Effect of a Patient-Centered Mobile App Self-Management Program for Osteoarthritis
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Chang Gung Memorial Hospital (Other)
Collaborators: National Science and Technology Council (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: ChangGungMHOA
Record Dates: First submitted 2022-11-09; First posted 2022-12-02 (Actual); Last update posted 2022-12-14 (Actual); Status verified 2022-11

CONDITIONS: Osteoarthritis
Keywords: osteoarthritis; self-management; mobile app; self-efficacy
MeSH Terms: conditions — Osteoarthritis | interventions — dimethyl sulfone

STUDY DESIGN:
Intervention Model Description: In the third year, we will test a patient-needs mobile app SM program for OA by randomized controlled trial of 6 months' duration. The total 66 patients with OA will be recruited while the participant in orthopedics clinic of a hospital. The experimental group (N=33) will receive a mSM program, and the control group (N=33) will receive with the usual care only.
Who Masked: Care Provider, Outcomes Assessor
Masking Description: Single (Outcomes Assessor) The researcher who applied the intervention program and the researcher who collected the data was never the same.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- The mobile app self-management (mSM) program focusing on patients' needs in OA patients (Experimental): An individualized mobile app self-management (mSM) program for managing OA patients' physical behavioral problems was applied for the intervention group. The program was based on the self-efficacy theory and the four resources were incorporated to emphasize patients' knowledge, skill, and responsibility in managing their OA situations.
  Interventions: Behavioral: A mobile app self-management (mSM) program
- Control group for mSM program (No Intervention): The control group will receive with the usual care only and follow-up 6 months.

INTERVENTIONS:
Behavioral: A mobile app self-management (mSM) program — The mSM program is developed on Bundura's self-efficacy theory, which provides four sources of information for SM. The strategies of the mSM consist of mobile app to management program including peer support, appraisal, goal setting and self-monitoring of exercise for OA and symptom management.
  Arms: The mobile app self-management (mSM) program focusing on patients' needs in OA patients

SUMMARY:
Aim: The aim of this study is to develop and evaluate the efficacy of a mobile app self-management (mSM) program focusing on patients' needs in OA patients over a 6 months' follow-up.

Methods: This study will be conducted in three years. In the first year, a qualitative needs assessment will be conducted to explore 20 parents' needs for improvements of the SM program until the saturation is reached. The specific requirements of the mSM users based on the parents' needs will be identified. In the second year, after patients' needs identified, the mSM program focusing on patients' needs will be developed through the literature searched and experts consulted. The mSM program contents, prototype, mobile application, field usability, and user acceptance will be tested by a 4-month pilot study. To ensure the protocol is realistic and whether any modifications of the program procedure are required by running pilot study with 10 OA patients. In the third year, we will test a patient-needs mobile app SM program for OA by randomized controlled trial of 6 months' duration. The total 66 patients with OA will be recruited while the participant in orthopedics clinic of a hospital. The experimental group (N=33) will receive a mSM program, and the control group (N=33) will receive with the usual care only. In order to examine the effects of mSM program, data will be collected with 4 time points which will be conducted at baseline (pre-discharge hospital) and at 1, 3, and 6 months, and by seven health- related outcomes that include physical function, quality of OA care, self-efficacy, quality of life, SM behaviors, and health services use. Outcome measures of this study will be analyzed using descriptive and inferential statistics with the generalized estimating equations analysis.

DETAILED DESCRIPTION:
Background: Osteoarthritis (OA) is a progressively degenerative disease, and is a leading cause of disability with incidence and prevalence rising in most elderly populations which contribute the number of OA continue increasing at a rapid rate. Indeed, the symptoms of OA can cause disability, pain, and joint stiffness, even results poorer quality of life. Self-management (SM) is worldwide reported as an effective approach to utilize for those with chronic disease. However, we had been conducted a program that granted by the Ministry of Science and Technology (NSC 102-2628-B-182-019-MY3), which showed the traditional SM program have some limitation such as patients can't get help immediately, follow up the patients' needs, fraud issue, involving all patients because geographical barriers, and the effectiveness don't remain long term. Therefore, it is need to develop of scalable eHealth SM models and practices seems mandatory in order to cope with the change in population needs and reduce the burden of OA. Aim: The aim of this study is to develop and evaluate the efficacy of a mobile app self-management (mSM) program focusing on patients' needs in OA patients over a 6 months' follow-up.

Methods: This study will be conducted in three years. In the first year, a qualitative needs assessment will be conducted to explore 20 parents' needs for improvements of the SM program until the saturation is reached. The specific requirements of the mSM users based on the parents' needs will be identified. In the second year, after patients' needs identified, the mSM program focusing on patients' needs will be developed through the literature searched and experts consulted. The mSM program contents, prototype, mobile application, field usability, and user acceptance will be tested by a 4-month pilot study. To ensure the protocol is realistic and whether any modifications of the program procedure are required by running pilot study with 10 OA patients. In the third year, we will test a patient-needs mobile app SM program for OA by randomized controlled trial of 6 months' duration. The total 66 patients with OA will be recruited while the participant in orthopedics clinic of a hospital. The experimental group (N=33) will receive a mSM program, and the control group (N=33) will receive with the usual care only. The mSM program is developed on Bundura's self-efficacy theory, which provides four sources of information for SM. The strategies of the mSM consist of mobile app to management program including peer support, appraisal, goal setting and self-monitoring of exercise for OA and symptom management. In order to examine the effects of mSM program, data will be collected with 4 time points which will be conducted at baseline (pre-discharge hospital) and at 1, 3, and 6 months, and by seven health- related outcomes that include physical function, quality of OA care, self-efficacy, quality of life, SM behaviors, and health services use. Outcome measures of this study will be analyzed using descriptive and inferential statistics with the generalized estimating equations analysis.

ELIGIBILITY:
Inclusion Criteria:

* Participants aged 45 years more with primary or secondary diagnosis of OA
* At a clinically stable with no signs of disease exacerbation in the last 30 days
* Ability to use and learn app for mobile phone

Exclusion Criteria:

* With severe comorbidities such as metastatic disease, pathological fractures, infection, or acute trauma
* Unstable physical and terminal illnesses
* Severe cognitive impairments or another debilitating psychiatric disorder
* Contraindication to physical activity such as walking
* Participation in another research protocol

Min Age: 45 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 66 (Estimated)
Dates: Start 2019-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-07-31 (Estimated)

PRIMARY OUTCOMES:
OsteoArthritis Quality Indicator (OA-QI) questionnaire version 2 (v2) | 6 months
  The OA-QI v2 is a joint specific outcome measure tool designed to assess patient-reported quality of OA care and to provide quality indicator in pass rates. Each item has three response option with 'Yes', 'No' and a third response which item is not applicable (for example, 'Not overweight' for the items on weight management) or the participant do not remember in 16 QI items. Scoring involves summating the total for each item score between 0-100, with a higher score indicating greater disability.
Arthritis Self-efficacy Scale (ASE) | 6 months
  The 11-items ASE scale is made up of two subscale including "ASE: Pain" and "ASE: Other Symptoms" will be used in current study. The research subjects will be asked to respond using a visual analogue scales (1-10) ranging from 1 "very uncertain", to 10 "very certain". Scores are summed across the items for each subscale to give a total score with a range of 5-50 for ASE- Pain (5 items), and 6-60 for ASE- Other Symptoms (6 items), with higher scores indicating higher confidence in arthritis self-efficacy.
Self-management behaviors scale | 6 months
  Cognitive symptom managements will assess using scales with each item rated in a six-point scale (0-5) anchored by "never" and "always". Scoring involves summating the total for each item score between 0-30, with a higher score indicating greater behaviors of self-management.

SECONDARY OUTCOMES:
EuroQol 5 Dimensions, European Quality of Life Five Dimension, and EuroQol five-dimensional. (EQ-5D-5L) | 6 months
  The EQ-5D-5L essentially consists of 2 pages: the EQ-5D descriptive system and the EQ visual analogue scale (VAS). The descriptive system comprises five dimensions: The patient is asked to indicate their health state by ticking the box next to the most appropriate statement in each of the five dimensions. This decision results in a 1-digit number that expresses the level selected for that dimension. The digits for the five dimensions can be combined into a 5-digit number that describes the patient's health state, for example, scoring 1 being the best score with no problem. A higher score in the EQ-5D-5L indicated better the quality of life. Moreover, the EQ visual analogue scale (VAS) is a measure of overall self-rated health status for TODAY. Scoring involves summating the total for each item score between 0-100, with a higher score indicating good their health.
Sit-to-stand. 30 second chair stand test | 6 months
  A test of sit-to-stand activity. Also a test of lower body strength and dynamic balance. On the signal to begin, start the stop watch. Count the total number of chair stands (up and down equals one stand) completed in 30 seconds. If a full stand has been completed at 30 seconds (i.e. standing fully erect or on the way down to the sitting position), then this final stand is counted in the total. If a person cannot stand even once then the score for the test is zero. The maximum number of chair stand repetitions possible in a 30 second period.
Walking short distances. 4x10m fast-paced walk test | 6 months
  A test of short distance walking activity. Scoring as below:
  * Timing starts on the signal to start at the start line and terminates once the participant crosses back over the start line after completing the 40 m (4x10 m).
  * When the participant crosses the 10m mark, timing is paused whilst the participant turns around the cone and then is resumed once they cross the 10m mark again. The same is repeated for the following turns and is stopped once the participant crosses the start line for the final time.
  * Time of one trial is recorded to the nearest 100th of a second.
  * Time of one test trial is recorded and expressed as speed m/s by dividing distance (40m) by time (s).
  * Regular walking aid is allowed and use should be recorded.
  * Minimal reporting standards: Assistive devices such as usual walking aids - walking stick et.
Health services use | 6 months
  Health services use will be measured from the self-reported number of contacts with a general physician, orthopedist, and other medical specialists including clinical and emergency visits as well as hospitalizations on all patients.

CONTACTS AND LOCATIONS:
Overall Officials: Junghua SHAO, Principal Investigator — Chang Gung Memorial Hospital
Locations (1):
- Chang Gung Memorial Hospital, Taoyuan District, Taiwan

IPD SHARING:
Plan to Share IPD: No
NO yet